CLINICAL TRIAL: NCT02345993
Title: Extra-fine Formoterol/Beclomethasone in the Treatment of Asthmatic Crisis
Brief Title: Extra-fine Formoterol/Beclomethasone in Asthmatic Crisis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Jose Luis Miguel, MD, MsC, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C40-14
Record Dates: First submitted 2015-01-14; First posted 2015-01-26 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Asthma; Asthmatic Crisis
Keywords: formoterol/beclomethasone in asthmatic crisis; asthmatic crisis treatment
MeSH Terms: conditions — Asthma; Status Asthmaticus | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extra fine Formoterol/Beclomethasone (Active Comparator): Group receiving the drug additional to standard treatment standard treatment consisting in: Albuterol 2.5 mg via nebulizer at baseline, 0, 20, 40 minutes + Systemic steroid (methylprednisolone 60 mg) at the moment of evaluation
  + formoterol/beclomethasone, 3 puffs administered via aerochamber at baseline (0), 20, 40 minutes
  Interventions: Drug: Extra fine Formoterol/Beclomethasone
- Placebo (Placebo Comparator): Group receiving placebo additional to standard treatment consisting in:
  Albuterol 2.5 mg via nebulizer at baseline (0), 20, 40 minutes + Systemic steroid (methylprednisolone 60 mg) at the moment of evaluation
  + Placebo, 3 puffs administered via aerochamber at baseline (0), 20, 40 minutes

INTERVENTIONS:
Drug: Extra fine Formoterol/Beclomethasone — standard treatment consisting in: Albuterol 2.5 mg via nebulizer at baseline (0), 20, 40 minutes + Systemic steroid (methylprednisolone 60 mg) at the moment of evaluation
  + formoterol/beclomethasone, 3 puffs administered via aerochamber at baseline (0), 20, 40, 60 minutes
  Other Names: Innovair
  Arms: Extra fine Formoterol/Beclomethasone

SUMMARY:
The purpose of this study is to determine whether extra fine formoterol/beclomethasona are more effective in the treatment of asthmatic crisis when added to conventional treatment compared with conventional treatment alone.

DETAILED DESCRIPTION:
Inhaled corticosteroids still the cornerstone in treatment of stable asthma, while bronchodilators and systemic steroids are in asthmatic crisis.

Asthmatic exacerbations are events occurring in the natural course of the disease, require a change in actual medication and they are associated with risks of complications producing important economic costs.

Some is known about non-genomic effects of inhaled corticosteroids, making possible, at least in theory, having a positive effect on treatment of a crisis. On the other hand, formoterol has been shown to have a rapid beginning of action (3 minutes), persisting its effect during 12 hours and it has been shown to be as effective as albuterol in the treatment of a crisis.

The development of extra-fine particles has allowed reaching more distal zones in the lungs producing more deposition of the drug, which as well decrease adverse effects are lesser doses of the drug are needed.

According to that, aims of this work is to determine whether extra-fine formoterol/beclomethasona are more effective in the treatment of asthmatic crisis when added to conventional treatment compared with conventional treatment in terms of pulmonary function, symptoms, inflammation markers and rates of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* previous asthma diagnosis by physician
* spirometry with quality grade A, B or C
* presenting with asthmatic crisis in emergency room

Exclusion Criteria:

* imminent respiratory arrest
* respiratory comorbidities (COPD, cystic fibrosis, interstitial lung disease, pneumothorax, bronchiectasis)
* use of systemic steroids in 3 months previous
* allergy to steroids
* Peripheral capillary oxygen saturation (SpO2) less than 88%.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function | 120 minutes
  change in Forced Expiratory Volume in 1 second (FEV1) with respect to basal

SECONDARY OUTCOMES:
Need for hospitalization | 120 minutes
Change in perception of dyspnea | 90 minutes
  change in Borg and Transitional Dyspnea Index
Biomarkers of inflammation | 120 minutes
  change in C- reactive protein, TNF-alpha, eosinophils
interleukins | 120 min
  change in eosinophilic and non eosinophilic interleukins (IL-4, IL-5, IL-13, IL-17, IL-33)

OTHER OUTCOMES:
Length of stay in hospital | 1 week
  in patients requiring hospitalisation, evaluate length of stay
adverse effects | 1 week
  adverse effects related to the drug

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Miguel, MD, MsC, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- National Institute of Respiratory Diseases, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Martinez FD, Vercelli D. Asthma. Lancet. 2013 Oct 19;382(9901):1360-72. doi: 10.1016/S0140-6736(13)61536-6. Epub 2013 Sep 13. PMID 24041942
- [Background] Garcia-Sancho C, Fernandez-Plata R, Martinez-Briseno D, Franco-Marina F, Perez-Padilla JR. [Adult asthma in Mexico City: a population-based study]. Salud Publica Mex. 2012 Jul-Aug;54(4):425-32. doi: 10.1590/s0036-36342012000400013. Spanish. PMID 22832835
- [Background] Rodrigo GJ, Rodrigo C, Hall JB. Acute asthma in adults: a review. Chest. 2004 Mar;125(3):1081-102. doi: 10.1378/chest.125.3.1081. PMID 15006973
- [Background] Lipworth B, Manoharan A, Anderson W. Unlocking the quiet zone: the small airway asthma phenotype. Lancet Respir Med. 2014 Jun;2(6):497-506. doi: 10.1016/S2213-2600(14)70103-1. PMID 24899370